CLINICAL TRIAL: NCT01199263
Title: A Randomized Phase II Evaluation of Weekly Paclitaxel (NSC# 673089) Versus Weekly Paclitaxel With Oncolytic Reovirus (Reolysin NSC # 729968) in the Treatment of Recurrent or Persistent Ovarian, Fallopian Tube or Primary Peritoneal Cancer
Brief Title: Paclitaxel With or Without Viral Therapy in Treating Patients With Recurrent or Persistent Ovarian Epithelial, Fallopian Tube, or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02654; NCI-2011-02654 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000684693; GOG-0186H (Other: NRG Oncology); GOG-0186H (Other: CTEP); U10CA180868 (NIH); U10CA027469 (NIH)
Record Dates: First submitted 2010-09-09; First posted 2010-09-10 (Estimated); Results first posted 2019-10-30 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-08

CONDITIONS: Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Paclitaxel; Taxes; reolysin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (paclitaxel) (Experimental): Patients receive paclitaxel IV over 1 hour on days 1, 8, and 15.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Paclitaxel
- Arm II (paclitaxel and wild-type reovirus) (Experimental): Patients receive paclitaxel as in arm I and wild-type reovirus IV over 1 hour on days 1-5.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Biological: Pelareorep

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Biological: Pelareorep — Given IV
  Other Names: PO BB0209; PO-BB0209; Reolysin; Reovirus Serotype 3; Wild-type Reovirus
  Arms: Arm II (paclitaxel and wild-type reovirus)

SUMMARY:
This randomized phase II trial studies the side effects and how well giving paclitaxel with or without viral therapy works in treating patients with ovarian epithelial, fallopian tube, or primary peritoneal cancer that has come back. Drugs used in chemotherapy, such as paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them spreading. Viral therapy may be able to kill tumor cells without damaging normal cells. Giving paclitaxel together with viral therapy may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the progression-free survival hazard ratio of the combination of weekly paclitaxel with Reolysin (wild-type reovirus) to weekly paclitaxel alone in patients with persistent or recurrent ovarian, fallopian tube, or primary peritoneal cancer.

II. To determine the frequency and severity of adverse events associated with treatment with weekly paclitaxel alone and weekly paclitaxel with REOLYSIN as assessed by Common Terminology Criteria for Adverse Events (CTCAE).

SECONDARY OBJECTIVES:

I. To estimate the progression-free survival and overall survival of patients treated with weekly paclitaxel alone and weekly paclitaxel with REOLYSIN.

II. To estimate (and compare) the proportion of patients who respond to the regimen on each arm of the study (according to Response Evaluation Criteria in Solid Tumors [RECIST] 1.1 with measurable patients and by cancer antigen [CA]-125 for those patients with detectable disease only).

III. To characterize and compare progression-free survival and overall survival in patients with measurable disease (RECIST 1.1 criteria) and patients with detectable (non-measurable) disease.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive paclitaxel intravenously (IV) over 1 hour on days 1, 8, and 15.

ARM II: Patients receive paclitaxel as in arm I and wild-type reovirus IV over 1 hour on days 1-5.

In both arms, treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have recurrent or persistent epithelial ovarian, fallopian tube or primary peritoneal carcinoma; histologic documentation of the original primary tumor is required via the pathology report
* Patients must have measurable disease or detectable (non-measurable) disease:

  * Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded); each lesion must be >= 10 mm when measured by computed tomography [CT], magnetic resonance imaging [MRI] or caliper measurement by clinical exam; or >= 20 mm when measured by chest x-ray; lymph nodes must be > 15 mm in short axis when measured by CT or MRI
  * Detectable (non-measurable) disease is defined as not having measurable disease but has at least one of the following conditions:

    * Baseline values of CA-125 at least 2 x upper limit of normal (ULN);
    * Ascites and/or pleural effusion attributed to tumor;
    * Solid and/or cystic abnormalities on radiographic imaging that do not meet RECIST 1.1 definitions for target lesions
* Patient with measurable disease must have at least one "target lesion" to be used to assess response on this protocol as defined by RECIST 1.1; tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days following completion of radiation therapy
* Patients must not be eligible for a higher priority Gynecologic Oncology Group (GOG) protocol, if one exists; in general, this would refer to any active GOG phase III protocol or rare tumor protocol for the same patient population
* Patients who have received one prior regimen must have a GOG performance status of 0, 1, or 2

  * Patients who have received two or three prior regimens must have a GOG performance status of 0 or 1
* Recovery from effects of recent surgery, radiotherapy, or chemotherapy:

  * Patients should be free of active infection requiring antibiotics (with the exception of uncomplicated urinary tract infection [UTI])
  * Any hormonal therapy directed at the malignant tumor must be discontinued at least one week prior to registration; continuation of hormone replacement therapy is permitted
  * Any other prior therapy directed at the malignant tumor, including chemotherapy, biologic/targeted and immunologic agents, must be discontinued at least three weeks prior to registration
* Patients must have had one prior platinum-based chemotherapeutic regimen for management of primary disease containing carboplatin, cisplatin, or another organoplatinum compound; this initial treatment may have included intraperitoneal therapy, consolidation, non-cytotoxic agents (biologic/targeted) or extended therapy administered after surgical or non-surgical assessment; if patients were treated with paclitaxel for their primary disease, this can have been given weekly or every 3 weeks
* Patients are allowed to receive, but are not required to receive, two additional cytotoxic regimens for management of recurrent or persistent disease, with no more than 1 non-platinum, non-taxane regimen; treatment with weekly paclitaxel for recurrent or persistent disease is NOT allowed
* Patients are allowed to receive, but are not required to receive, non-cytotoxic (biologic/targeted) therapy as part of their primary treatment regimen; patients are allowed to receive, but are not required to receive, non-cytotoxic (biologic/targeted) therapy as part of their treatment for recurrent or persistent disease and/or as treatment for recurrent or persistent disease; if non-cytotoxic (biologic/targeted) therapy is given alone (i.e., not in combination with cytotoxic chemotherapy) it will NOT count as a prior regimen

  * For the purposes of this study, poly (adenosine diphosphate [ADP]-ribose) polymerase (PARP) inhibitors will NOT count as a prior regimen when given alone (i.e., not in combination with cytotoxic chemotherapy)
* Patients who have received only one prior cytotoxic regimen (platinum-based regimen for management of primary disease), must have a platinum-free interval of less than 12 months, or have progressed during platinum-based therapy, or have persistent disease after a platinum-based therapy
* Absolute neutrophil count (ANC) greater than or equal to 1,500/mcl
* Platelets greater than or equal to 100,000/mcl
* Hemoglobin greater than or equal to 9 g/dL
* Creatinine less than or equal to 1.5 x institutional upper limit normal (ULN)
* Bilirubin less than or equal to 1.5 x ULN
* Serum glutamic oxaloacetic transaminase (SGOT) less than or equal to 3 x ULN
* Alkaline phosphatase less than or equal to 2.5 x ULN
* Neuropathy (sensory and motor) less than or equal to grade 1
* Patients of childbearing potential must have a negative pregnancy test prior to the study entry and be practicing an effective form of contraception; (pregnant women are excluded from this study)
* Patients must have signed an approved informed consent and authorization permitting the release of personal health information
* Patients must meet pre-entry requirements as specified
* Patients must be able to avoid direct contact with severely immune-compromised individuals such as patients who have had a recent bone-marrow or organ transplant or patients with acquire immunodeficiency syndrome (AIDS); contact should be avoided on the days of Reolysin treatment and for the 2 days following Reolysin treatment
* Patients must be able to avoid direct contact with pregnant or nursing women and infants while receiving Reolysin; contact should be avoided on the days of Reolysin treatment and for the 2 days following Reolysin treatment

Exclusion Criteria:

* Patient who have had previous treatment with Reolysin or other oncolytic virus; patients who have had previous treatment with weekly paclitaxel for recurrent or persistent disease
* Patients with a history of other invasive malignancies, with the exception of non-melanoma skin cancer and other specific malignancies are excluded if there is any evidence of other malignancy being present within the last three years; patients are also excluded if their previous cancer treatment contraindicates this protocol therapy
* Patients who have received prior radiotherapy to any portion of the abdominal cavity or pelvis OTHER THAN for the treatment of ovarian, fallopian tube, or primary peritoneal cancer within the last three years are excluded; prior radiation for localized cancer of the breast, head and neck, or skin is permitted, provided that it was completed more than three years prior to registration, and the patient remains free of recurrent or metastatic disease
* Patients who have received prior chemotherapy for any abdominal or pelvic tumor OTHER THAN for the treatment of ovarian, fallopian tube, or primary peritoneal cancer within the last three years are excluded; patients may have received prior adjuvant chemotherapy for localized breast cancer, provided that it was completed more than three years prior to registration, and the patient remains free of recurrent or metastatic disease
* Patients with a past history of primary endometrial cancer are excluded unless all of the following conditions are met: stage not greater than I-B; no more than superficial myometrial invasion, without vascular or lymphatic invasion; no poorly differentiated subtypes, including papillary serious, clear cell or other International Federation of Gynecology and Obstetrics (FIGO) grade 3 lesions
* Patients with known human immunodeficiency virus (HIV) or hepatitis B or C are excluded due to risk of viral infectivity of Reolysin therefore patients with a pre-existent infection are not eligible
* Patients who are receiving immunosuppressive therapy including chronic oral steroids (at an equivalent dose of greater than prednisone 5 mg daily)
* Women who are pregnant or nursing; pregnant women are excluded from this study; breastfeeding should be discontinued while the mother is being treated with the agents in this clinical trial
* Myocardial infarction or unstable angina within 6 months of the first date of study therapy
* History of serious ventricular arrhythmia (i.e., ventricular tachycardia or ventricular fibrillation) or cardiac arrhythmias requiring anti-arrhythmic medications (except for atrial fibrillation that is well controlled with antiarrhythmic medication)
* Troponin > ULN
* Baseline ejection fraction < 50% as assessed by echocardiogram or multi gated acquisition scan (MUGA)
* New York Heart Association (NYHA) class II or greater congestive heart failure
* History of cerebrovascular accident (CVA, stroke), transient ischemic attack (TIA) or subarachnoid hemorrhage within six months of the first date of study therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2010-12-06 (Actual); Primary Completion 2015-06-01 (Actual); Study Completion 2020-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David E Cohn, Principal Investigator — NRG Oncology
Locations (36):
- United States (36):
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Beaumont Hospital - Dearborn, Dearborn, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Allegiance Health, Jackson, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Atrium Health Cabarrus/LCI-Concord, Concord, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Women and Infants Hospital, Providence, Rhode Island
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Carilion Clinic Gynecological Oncology, Roanoke, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Paclitaxel): Patients receive paclitaxel IV over 1 hour on days 1, 8, and 15. Laboratory Biomarker Analysis: Correlative studies Paclitaxel: Given IV
- Arm II (Paclitaxel and Wild-type Reovirus): Patients receive paclitaxel as in arm I and wild-type reovirus IV over 1 hour on days 1-5.
  Laboratory Biomarker Analysis: Correlative studies Paclitaxel: Given IV Pelareorep: Given IV
Period: Overall Study
Arm/Group | Arm I (Paclitaxel) | Arm II (Paclitaxel and Wild-type Reovirus)
Started | 54 | 54
Completed | 48 | 52
Not Completed | 6 | 2
Not completed — Ineligible | 0 | 2
Not completed — Never Treated | 6 | 0

BASELINE CHARACTERISTICS:
Population: All Enrolled participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Paclitaxel) | Arm II (Paclitaxel and Wild-type Reovirus) | Total
Number analyzed (Participants) | 54 | 54 | 108
Age, Customized [Count of Participants; unit: Participants]
  30-39 years | 1 | 0 | 1
  40-49 years | 4 | 4 | 8
  50-59 years | 19 | 11 | 30
  60-69 years | 20 | 26 | 46
  70-79 years | 9 | 11 | 20
  >=80 years | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 54 | 108
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 51 | 50 | 101
  Unknown or Not Reported | 0 | 4 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 50 | 48 | 98
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Time from patient entry until progression, death, or date last seen. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: Approximately 4.5 years.
Population: Enrolled patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm I (Paclitaxel) | Arm II (Paclitaxel and Wild-type Reovirus)
Number analyzed (Participants) | 54 | 54
Months | 3.94 [2.86 to 7.89] | 4.39 [2.60 to 5.52]

2. Primary Outcome: Number of Participants With Adverse Events Grade 3 or Greater as Assessed by CTCAE Version 4.0
Description: The frequency and severity of Grade 3 and above toxicities are tabulated.
Time Frame: approximately 4.5 years
Population: Eligible and treated participants
Measure: Count of Participants; unit: Participants
Groups:
- Arm I (Paclitaxel) Grade 3 and Above Toxicity: Grade 3 and above toxicity in patients who receive paclitaxel IV over 1 hour on days 1, 8, and 15.
- Arm II (Paclitaxel and Wild-type Reovirus) Grade 3 Above: Grade 3 and above toxicity in patients who receive paclitaxel as in arm I and wild-type reovirus IV over 1 hour on days 1-5.
Arm/Group | Arm I (Paclitaxel) Grade 3 and Above Toxicity | Arm II (Paclitaxel and Wild-type Reovirus) Grade 3 Above
Number analyzed (Participants) | 48 | 52
Participants
  Leukopenia | 3 | 17
  Thrombocytopenia | 0 | 1
  Neutropenia | 5 | 15
  Anemia | 7 | 10
  Other Investigations | 4 | 4
  Other Blood/lymphatics | 1 | 1
  Cardiac | 0 | 4
  Ear and Labyrinth | 1 | 0
  Eye | 1 | 0
  Nausea | 4 | 3
  Vomiting | 4 | 1
  Other gastrointestinal | 18 | 16
  General and administration site | 5 | 13
  Hepatobiliary | 0 | 2
  Infections/infestations | 5 | 7
  Injury/poisoning | 0 | 1
  Metabolism/nutrition | 11 | 11
  Musculoskeletal/connective tissue | 2 | 1
  Neoplasms benign/malignant | 1 | 5
  Peripheral sensory neuropathy | 1 | 0
  Nervous System | 2 | 6
  Renal/urinary | 2 | 2
  Reproductive/breast | 0 | 1
  Respiratory/thoracic/mediastinal | 1 | 13
  Vascular disorders | 11 | 15

3. Secondary Outcome: Percentage of Participants withTumor Response by RECIST
Description: Participants with Complete and Partial Tumor Response by RECIST. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: approximately 4.5 years
Population: All enrolled patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (Paclitaxel) | Arm II (Paclitaxel and Wild-type Reovirus)
Number analyzed (Participants) | 54 | 54
percentage of participants | 16.7 [7.9 to 29.3] | 13.0 [5.4 to 24.9]

4. Secondary Outcome: Median Overall Survival (OS) by Treatment Group
Description: Time from patient randomization to death or date last seen.
Time Frame: After patient stops protocol therapy, she is followed quarterly for 2 years, semi-annually for 3 more years, approximately 4.5 years.
Population: Enrolled patients.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm I (Paclitaxel) | Arm II (Paclitaxel and Wild-type Reovirus)
Number analyzed (Participants) | 54 | 54
Months | 13.1 [7.9 to 21.4] | 12.6 [8.2 to 18.2]

5. Secondary Outcome: Tumor Response by CA125
Description: Percentage of participants with Complete and Partial Tumor Response by CA125.
Time Frame: Before every cycle, approximately 4.5 years.
Population: All enrolled patients.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (Paclitaxel) | Arm II (Paclitaxel and Wild-type Reovirus)
Number analyzed (Participants) | 54 | 54
percentage of participants | 18.5 [9.3 to 31.4] | 22.2 [12.0 to 35.6]

ADVERSE EVENTS:
Time Frame: During study treatment (an average of 12 weeks) and up to 30 days after.
Arm/Group | Arm I (Paclitaxel) | Arm II (Paclitaxel and Wild-type Reovirus)
Serious Adverse Events (participants affected / at risk) | 17/48 | 24/52
Other Adverse Events (participants affected / at risk) | 48/48 | 52/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Paclitaxel) (N=48) | Arm II (Paclitaxel and Wild-type Reovirus) (N=52)
Anemia (Blood and lymphatic system disorders) | 0 | 2
Colonic Perforation (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 6 | 4
Abdominal Pain (Gastrointestinal disorders) | 1 | 0
Intra-Abdominal Hemorrhage (Gastrointestinal disorders) | 0 | 2
Esophagitis (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 2
Gastritis (Gastrointestinal disorders) | 0 | 1
Non-Cardiac Chest Pain (General disorders) | 0 | 1
Infusion Related Reaction (General disorders) | 0 | 1
Stoma Site Infection (Infections and infestations) | 1 | 0
Skin Infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Lung Infection (Infections and infestations) | 1 | 2
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 1
Creatinine Increased (Investigations) | 0 | 1
Neutrophil Count Decreased (Investigations) | 0 | 3
Blood Bilirubin Increased (Investigations) | 0 | 1
White Blood Cell Decreased (Investigations) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Neoplasms Benign, Malignant And Unspecified (Incl (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 5
Intracranial Hemorrhage (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 1 | 1
Vaginal Hemorrhage (Reproductive system and breast disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Thromboembolic Event (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Paclitaxel) (N=48) | Arm II (Paclitaxel and Wild-type Reovirus) (N=52)
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 43 | 48
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 0 | 5
Ventricular Tachycardia (Cardiac disorders) | 0 | 1
Sinus Bradycardia (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 3 | 2
Myocardial Infarction (Cardiac disorders) | 0 | 1
Acute Coronary Syndrome (Cardiac disorders) | 1 | 0
Sinus Tachycardia (Cardiac disorders) | 2 | 5
Chest Pain - Cardiac (Cardiac disorders) | 2 | 2
Tinnitus (Ear and labyrinth disorders) | 6 | 2
Hearing Impaired (Ear and labyrinth disorders) | 3 | 0
Ear Pain (Ear and labyrinth disorders) | 4 | 2
Adrenal Insufficiency (Endocrine disorders) | 0 | 1
Watering Eyes (Eye disorders) | 0 | 1
Flashing Lights (Eye disorders) | 1 | 2
Eye Pain (Eye disorders) | 2 | 0
Cataract (Eye disorders) | 2 | 1
Conjunctivitis (Eye disorders) | 1 | 0
Retinopathy (Eye disorders) | 0 | 1
Blurred Vision (Eye disorders) | 7 | 6
Floaters (Eye disorders) | 1 | 1
Extraocular Muscle Paresis (Eye disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 4
Dyspepsia (Gastrointestinal disorders) | 6 | 1
Dry Mouth (Gastrointestinal disorders) | 2 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 28 | 37
Diarrhea (Gastrointestinal disorders) | 20 | 27
Vomiting (Gastrointestinal disorders) | 20 | 24
Upper Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 0 | 1
Bloating (Gastrointestinal disorders) | 10 | 10
Stomach Pain (Gastrointestinal disorders) | 0 | 3
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0
Rectal Mucositis (Gastrointestinal disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 23 | 24
Rectal Hemorrhage (Gastrointestinal disorders) | 2 | 1
Mucositis Oral (Gastrointestinal disorders) | 10 | 16
Oral Hemorrhage (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Gastric Hemorrhage (Gastrointestinal disorders) | 1 | 0
Oral Pain (Gastrointestinal disorders) | 1 | 1
Abdominal Distension (Gastrointestinal disorders) | 7 | 5
Nausea (Gastrointestinal disorders) | 35 | 44
Gastroparesis (Gastrointestinal disorders) | 0 | 1
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 2 | 2
Rectal Pain (Gastrointestinal disorders) | 1 | 0
Esophagitis (Gastrointestinal disorders) | 2 | 0
Fecal Incontinence (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 5 | 5
Toothache (Gastrointestinal disorders) | 2 | 0
Anal Fistula (Gastrointestinal disorders) | 0 | 1
Esophageal Pain (Gastrointestinal disorders) | 2 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1
Esophageal Hemorrhage (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 2 | 1
Pain (General disorders) | 9 | 21
Malaise (General disorders) | 1 | 2
Localized Edema (General disorders) | 5 | 3
Injection Site Reaction (General disorders) | 0 | 1
Infusion Site Extravasation (General disorders) | 0 | 1
Flu Like Symptoms (General disorders) | 2 | 18
Edema Trunk (General disorders) | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 6 | 8
Edema Limbs (General disorders) | 18 | 15
Facial Pain (General disorders) | 1 | 0
Edema Face (General disorders) | 1 | 3
Fatigue (General disorders) | 40 | 44
Fever (General disorders) | 7 | 27
Gait Disturbance (General disorders) | 0 | 1
Chills (General disorders) | 4 | 33
Infusion Related Reaction (General disorders) | 1 | 2
Hepatobiliary Disorders - Other (Hepatobiliary disorders) | 0 | 1
Gallbladder Pain (Hepatobiliary disorders) | 0 | 1
Gallbladder Obstruction (Hepatobiliary disorders) | 0 | 1
Allergic Reaction (Immune system disorders) | 2 | 2
Wound Infection (Infections and infestations) | 0 | 1
Upper Respiratory Infection (Infections and infestations) | 2 | 2
Soft Tissue Infection (Infections and infestations) | 1 | 0
Skin Infection (Infections and infestations) | 2 | 2
Sinusitis (Infections and infestations) | 2 | 5
Sepsis (Infections and infestations) | 2 | 1
Salivary Gland Infection (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Peritoneal Infection (Infections and infestations) | 1 | 0
Otitis Media (Infections and infestations) | 1 | 0
Papulopustular Rash (Infections and infestations) | 1 | 0
Nail Infection (Infections and infestations) | 0 | 1
Mucosal Infection (Infections and infestations) | 0 | 1
Lung Infection (Infections and infestations) | 1 | 2
Laryngitis (Infections and infestations) | 0 | 1
Esophageal Infection (Infections and infestations) | 1 | 0
Conjunctivitis Infective (Infections and infestations) | 0 | 1
Gum Infection (Infections and infestations) | 0 | 1
Vaginal Infection (Infections and infestations) | 0 | 3
Urinary Tract Infection (Infections and infestations) | 13 | 11
Bronchial Infection (Infections and infestations) | 1 | 0
Enterocolitis Infectious (Infections and infestations) | 0 | 3
Bladder Infection (Infections and infestations) | 0 | 1
Postoperative Hemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 1
Burn (Injury, poisoning and procedural complications) | 0 | 1
Bruising (Injury, poisoning and procedural complications) | 2 | 1
Weight Loss (Investigations) | 4 | 4
Weight Gain (Investigations) | 4 | 3
Platelet Count Decreased (Investigations) | 11 | 30
Lymphocyte Count Decreased (Investigations) | 6 | 4
Inr Increased (Investigations) | 2 | 3
Creatinine Increased (Investigations) | 13 | 14
Cholesterol High (Investigations) | 1 | 0
Neutrophil Count Decreased (Investigations) | 25 | 39
Urine Output Decreased (Investigations) | 1 | 0
Blood Bilirubin Increased (Investigations) | 3 | 3
White Blood Cell Decreased (Investigations) | 35 | 42
Aspartate Aminotransferase Increased (Investigations) | 11 | 8
Alkaline Phosphatase Increased (Investigations) | 9 | 8
Alanine Aminotransferase Increased (Investigations) | 7 | 6
Activated Partial Thromboplastin Time Prolonged (Investigations) | 4 | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 3 | 5
Hyponatremia (Metabolism and nutrition disorders) | 15 | 15
Hypomagnesemia (Metabolism and nutrition disorders) | 11 | 14
Hypokalemia (Metabolism and nutrition disorders) | 10 | 9
Hypoglycemia (Metabolism and nutrition disorders) | 3 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 16 | 16
Hypoalbuminemia (Metabolism and nutrition disorders) | 21 | 25
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 0
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 | 0
Hypernatremia (Metabolism and nutrition disorders) | 4 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 2 | 4
Hyperkalemia (Metabolism and nutrition disorders) | 3 | 5
Hyperglycemia (Metabolism and nutrition disorders) | 17 | 19
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 9 | 7
Anorexia (Metabolism and nutrition disorders) | 22 | 27
Acidosis (Metabolism and nutrition disorders) | 1 | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 6 | 7
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 13
Muscle Weakness Lower Limb (Musculoskeletal and connective tissue disorders) | 1 | 1
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 9 | 10
Flank Pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 4 | 2
Bone Pain (Musculoskeletal and connective tissue disorders) | 8 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 8 | 15
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 | 10
Tremor (Nervous system disorders) | 2 | 0
Presyncope (Nervous system disorders) | 0 | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 30 | 33
Peripheral Motor Neuropathy (Nervous system disorders) | 2 | 2
Paresthesia (Nervous system disorders) | 0 | 1
Memory Impairment (Nervous system disorders) | 2 | 0
Lethargy (Nervous system disorders) | 0 | 1
Movements Involuntary (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 11 | 19
Facial Muscle Weakness (Nervous system disorders) | 0 | 1
Dysphasia (Nervous system disorders) | 2 | 0
Dysgeusia (Nervous system disorders) | 4 | 3
Sinus Pain (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 2
Dizziness (Nervous system disorders) | 9 | 12
Depressed Level Of Consciousness (Nervous system disorders) | 0 | 1
Cognitive Disturbance (Nervous system disorders) | 2 | 1
Ataxia (Nervous system disorders) | 0 | 1
Akathisia (Nervous system disorders) | 1 | 1
Suicidal Ideation (Psychiatric disorders) | 0 | 1
Restlessness (Psychiatric disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 11 | 12
Depression (Psychiatric disorders) | 18 | 16
Confusion (Psychiatric disorders) | 2 | 2
Anxiety (Psychiatric disorders) | 10 | 11
Agitation (Psychiatric disorders) | 1 | 1
Urinary Urgency (Renal and urinary disorders) | 5 | 1
Urinary Tract Obstruction (Renal and urinary disorders) | 1 | 1
Urinary Retention (Renal and urinary disorders) | 2 | 0
Urinary Incontinence (Renal and urinary disorders) | 4 | 4
Urinary Tract Pain (Renal and urinary disorders) | 5 | 6
Urinary Frequency (Renal and urinary disorders) | 8 | 9
Proteinuria (Renal and urinary disorders) | 3 | 0
Hematuria (Renal and urinary disorders) | 2 | 3
Chronic Kidney Disease (Renal and urinary disorders) | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 1 | 2
Vaginal Pain (Reproductive system and breast disorders) | 0 | 1
Vaginal Hemorrhage (Reproductive system and breast disorders) | 2 | 0
Vaginal Dryness (Reproductive system and breast disorders) | 1 | 0
Pelvic Pain (Reproductive system and breast disorders) | 1 | 1
Vaginal Discharge (Reproductive system and breast disorders) | 1 | 0
Breast Pain (Reproductive system and breast disorders) | 1 | 0
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinus Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 7 | 10
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 5
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Sleep Apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 7
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 24 | 30
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 18
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Skin And Subcutaneous Tissue Disorders - Other (Skin and subcutaneous tissue disorders) | 0 | 1
Rash Acneiform (Skin and subcutaneous tissue disorders) | 2 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 8
Palmar-Plantar Erythrodysesthesia Syndrome (Skin and subcutaneous tissue disorders) | 1 | 1
Pain Of Skin (Skin and subcutaneous tissue disorders) | 0 | 1
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 10 | 6
Nail Ridging (Skin and subcutaneous tissue disorders) | 1 | 1
Nail Loss (Skin and subcutaneous tissue disorders) | 4 | 5
Nail Discoloration (Skin and subcutaneous tissue disorders) | 5 | 5
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 0 | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 2 | 5
Bullous Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 35 | 36
Thromboembolic Event (Vascular disorders) | 4 | 4
Superficial Thrombophlebitis (Vascular disorders) | 0 | 1
Lymphedema (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 6 | 7
Hypertension (Vascular disorders) | 15 | 20
Hot Flashes (Vascular disorders) | 10 | 7
Flushing (Vascular disorders) | 4 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less